CLINICAL TRIAL: NCT02767167
Title: Contribution of Cow's Milk to Iodine and Selenium Status in Women of Child-bearing Age
Acronym: SIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Dairy Council for Northern Ireland (Other); LGC Limited (Industry); University Hospital Southampton NHS Foundation Trust (Other); Northern Health and Social Care Trust (Other Government); Department of Agriculture and Rural Development Northern Ireland (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/15/0042
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-04

CONDITIONS: Selenium and Iodine Status
Keywords: Cow's milk; Iodine; Selenium; Women; Child-bearing age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milk treatment group (Active Comparator): Semi-skimmed cow's milk + normal diet for 12 weeks
  Interventions: Other: Semi-skimmed cow's milk
- Control group (No Intervention): Normal diet for 12 weeks

INTERVENTIONS:
Other: Semi-skimmed cow's milk — 430ml of semi-skimmed cow's milk / day for 12 weeks
  Arms: Milk treatment group

SUMMARY:
Iodine is an essential trace element necessary for the synthesis of thyroid hormones which are critical for human growth and development throughout the lifecycle. Iodine is particularly important during pregnancy and infancy for brain and neurological development. Severe iodine deficiency during pregnancy can cause severe mental impairment and stillbirth while mild-to-moderate deficiency has been associated with impaired infant development. As such, pregnant women and women of child-bearing age are particularly vulnerable to the effects of iodine deficiency.

Globally, 241 million (30%) school aged children are iodine deficient. Historically, the UK and Ireland were believed to be iodine sufficient but concern has been expressed in the last decade regarding the iodine status of the UK and Irish populations. A study of Irish women in 2004 reported 55% of pregnant women in their sample population to be moderately iodine deficient and 53% of non-pregnant women to be moderately iodine deficient. A study of UK schoolgirls found that 51% were mildly iodine deficient and 16% were moderately deficient. Importantly, the prevalence of iodine deficiency was highest in Northern Ireland where 85% of those sampled were iodine deficient.

Iodine is known to interact with selenium in the conversion of the thyroid hormone thyroxine (T4) to the metabolically active triiodothyonine (T3) hormone. Selenium is also important for immune, cardiovascular and cognitive function. Selenium status has been reported to be moderately low using pooled English data on blood selenium concentrations from 1984 to 1992. In addition, the latest National Diet and Nutrition Survey reports that selenium intakes are below recommendations for several population groups including women of childbearing age where mean selenium intakes are 76% of the recommended 60µg/day. This national survey also reported that 49% of women aged 19-64 years failed to meet the lower reference nutrient intake of 40µg/day.

Milk and dairy products are the major source of iodine for the UK population and are also a source of selenium. The contribution of milk and dairy products to iodine and selenium intakes is greatest in adult females (35% and 6% respectively). Observational evidence has repeatedly reported milk consumption to be positively correlated with iodine status and iodine intakes. Research in Iceland and New Zealand has reported that milk consumption is not associated with selenium status; however it is unknown if this is true for the UK population.

To date, no randomised controlled trial has examined the effect of milk consumption on either iodine or selenium status. The possibility of increasing iodine and selenium intake by increasing milk consumption, a widely available and consumed foodstuff, in a population group vulnerable to micronutrient deficiency should be investigated. This would add valuable data to the knowledge base for iodine, where there is ongoing debate over the most appropriate means of increasing iodine intake amongst women of childbearing age in the UK where salt iodisation, the key strategy in preventing deficiency, is not implemented.

The aim of this study is to investigate the impact of cow's milk consumption on the biological status of iodine and selenium among women of child-bearing age.

The study will be a 12 week randomised-controlled human intervention study. Participants will be randomised to consume additional semi-skimmed milk in the Following amounts, control group (0mls/day), intervention group (430mls/day or 3l per week).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Healthy
* Age 18-45 years
* Females
* Non smoking
* No history of thyroid or gastrointestinal conditions
* Not consuming thyroid medication or medication containing iodine or selenium
* Willing to increase their milk consumption should they be randomised into the milk group

Exclusion Criteria:

* Smoker
* Pregnant, breastfeeding or planning to become pregnant during the study
* Milk allergy
* Non-milk consumers or vegans
* Lactose intolerant individuals
* Use of dietary supplements containing iodine or selenium in previous 3 months
* Peri- or post-menopausal
* Consume more than 250ml of milk daily

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | Change from baseline following 12-week intervention

SECONDARY OUTCOMES:
Serum thyroid hormone analysis | Baseline (week 0), mid (week 6) and post-intervention (week 12)
Urinary creatinine analysis | Baseline (week 0), mid (week 6) and post-intervention (week 12)
Serum selenoprotein P analysis | Baseline (week 0), mid (week 6) and post-intervention (week 12)
Dietary iodine and selenium intake | Baseline (week 0), mid (week 6) and post-intervention (week 12)
  24-hour dietary recall
Blood pressure | Baseline (week 0), mid (week 6) and post-intervention (week 12)
Body Mass Index | Baseline (week 0), mid (week 6) and post-intervention (week 12)
Waist Hip ratio | Baseline (week 0), mid (week 6) and post-intervention (week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Kane SM, Pourshahidi LK, Mulhern MS, Strain JJ, Mackle EM, Koca D, Schomburg L, Hill S, O'Reilly J, Kmiotek D, Deitrich C, Bath SC, Yeates AJ. Cow Milk Consumption Increases Iodine Status in Women of Childbearing Age in a Randomized Controlled Trial. J Nutr. 2018 Mar 1;148(3):401-408. doi: 10.1093/jn/nxx043. PMID 29546298